CLINICAL TRIAL: NCT01715922
Title: Prospective Pilot Study to Evaluate a Standardized Management of Cryptococcal Meningitis in Patients Infected With HIV in Sub-Saharan Africa Involving an Initial Combination Therapy With Fluconazole and Flucytosine in High Doses, Complemented by Repeat Lumbar Punctures
Brief Title: Study Evaluating Efficiency and Tolerance of High-dose Fluconazole Associated With Flucytosine as Induction Therapy for Cryptococcal Meningitis Associated With HIV in Sub-saharan Africa
Acronym: Flucocrypto
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: CHU Kamenge, BURUNDI (Unknown); Hospital Avicenne (Other); Institut Pasteur (Industry); Hôpital Necker-Enfants Malades (Other); Institut de Médecine et Epidémiologie Appliquée (IMEA) (Unknown); Hôpital de Treichville (Unknown); Hôpital Cocody (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12257 Flucocrypto
Record Dates: First submitted 2012-10-19; First posted 2012-10-29 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Cryptococcal Meningitis; HIV
Keywords: Cryptococcal meningitis; HIV Infections; Oral treatment; High dose of fluconazole; Flucytosine; Burundi; Ivory Coast
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections | interventions — Fluconazole; Flucytosine; Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- oral treatment (Other): Drug: Fluconazole and flucytosine
  Induction treatment for 2 weeks:
  Fluconazole (1600mg/j) + flucytosine (100 mg/kg/j) lumbar punctures to control intracranial pressure Consolidation treatment for 8 weeks: fluconazole (800 mg/j)
  Interventions: Drug: Fluconazole; Drug: Flucytosine; Procedure: lumbar punctures

INTERVENTIONS:
Drug: Fluconazole — Induction treatment for 2 weeks: Fluconazole (1600mg/j) Consolidation treatment for 8 weeks: fluconazole (800 mg/j)
Drug: Flucytosine — Flucytosine (100 mg/kg/j) for 2 weeks
Procedure: lumbar punctures — lumbar punctures to control intracranial pressure

SUMMARY:
The aim of the trial is to demonstrate that in a sub-Saharan African setting, the association of:

1. Oral treatment : high dose of fluconazole (1600mg/d) associated with flucytosine (100 mg/kg/j) as induction therapy
2. lumbar punctures to control intracranial pressure

can decrease mortality rate below 35% at 10 weeks.

This is a non-randomized open label pilot study, with standardized management of cryptococcoses meningitis and follow-up in Burundi and Ivory Coast. A total of 41 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* HIV Infection
* First episode of cryptococcal meningitis on basis CSF India ink and/or CSF cryptococcal antigen.
* Glasgow > 9 after lumbar punctures
* Absence of peripheral focal deficit in the limbs
* informed consent signed

Exclusion Criteria:

* Hemoglobin <7.5 g / dl;
* neutrophils count <500/mm3;
* Platelets count <50 000/mm3;
* transaminases > 5 times upper limit of normal;
* Troubles with severe mental alertness Glasgow <9 after the initial lumbar puncture;
* focal neurological deficit in the limbs;
* Pregnancy or lactation on going;
* Ongoing systemic antifungal treatment;
* History of cryptococcal meningitis;
* Ongoing rifampicin and ritonavir treatment;
* Subject participating in another study with a risk of mutual interference on the interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-05; Primary Completion 2015-09 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | 10 weeks

SECONDARY OUTCOMES:
Mortality rate | 14 days and 24 weeks
Percentage of patients with negative cerebrospinal fluid (CSF) cultures | 14 days and 10 weeks
Number of relapses of cryptococcal throughout the monitoring period | up to 24 weeks
Number of "Immune Reconstitution Inflammatory Syndrome" (IRIS) throughout the monitoring period | up to 24 weeks
  The IRIS diagnosis criteria will be those given in: Bicanic T, et al. Immune Reconstitution Inflammatory Syndrome in HIV-associated cryptococcal meningitis: a prospective study, J Acquir Immune Defic Syndr 2009; 51:130-134.
Number and severity of adverse events | up to 24 weeks
Cerebrospinal fluid pressure evolution | up to 24 weeks
Percentage of patients with undetectable viral load | 24 weeks
CD4 count | 24 weeks
Concentration of flucytosine in cerebrospinal fluid | 28 days or 10 weeks
Sensitivity of cryptococcal antigen by strip method LFA (lateral-flow immunoassay) | at study entry
  on urines, plasma, CSF and whole blood fingerstick
CSF total volume discharged | up to 24 weeks
Number of lumbar punctures performed | up to 24 weeks
Concentration of fluconazole in plasma | 28 days or 10 weeks
Concentration of fluconazole in cerebrospinal fluid | 28 days or 10 weeks
Concentration of flucytosine in plasma | 28 days or 10 weeks
MICs of fluconazole | 28 days
  MICs of fluconazole for cryptococcus strains, if CSF cultures ar positive at 28 days or 10 weeks or in case of relapse

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Bouchaud, PhD, Study Chair — Hopital Avicenne, Service des maladies infectieuses, Paris, france; Théodore Niyangobo, PhD, Study Chair — CHU Kamenge, Bujumbura, Burundi; Amélie Chabrol, MD, Principal Investigator — Hopital Avicenne, Service des maladies infectieuses, Paris, france; Kakou AKA, Professor, Principal Investigator — CHU Triechville
Locations (7):
- Burundi (5):
  - CHU Kamenge, Bujumbura
  - Hôpital Prince Régent Charles, Bujumbura
  - Hôpital général, Bururi
  - Hôpital général, Kayanza
  - Hôpital général, Muyinga
- Côte d’Ivoire (2):
  - Service de Maladies Infectieuses & Tropicales - Hôpital Triechville, Abidjan
  - Service de Neurologie - Hôpital Cocody, Abidjan

REFERENCES:
- See also: Sponsor web page — http://www.anrs.fr